CLINICAL TRIAL: NCT04662632
Title: A Randomized Controlled Trial of Alternating Irrigation of Vancomycin Hydrochloride and Tobramycin Sulfate in Patients Undergoing Two-Stage Exchange Arthroplasty for Periprosthetic Joint Infection (PJI) of the Hip or Knee
Brief Title: Abbreviated Protocol for Two-Stage Exchange
Acronym: APEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Osteal Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JPS-0301
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Prosthetic Joint Infection
Keywords: Hip; Knee; Biofilm; Minimum-biofilm-eradication-concentration
MeSH Terms: interventions — Tobramycin; Standard of Care; Vancomycin

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded to their randomization arm assignment until the completion of Stage 1 surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Experimental (Experimental): Local antibiotic irrigation via the VT-X7 (Vancomycin and Tobramycin Exchanged over 7 Days) Treatment System adjuvant to two-stage exchange arthroplasty per standard of care.
  Interventions: Combination Product: VT-X7 Treatment System with Tobramycin Sulfate; Procedure: Two-stage exchange arthroplasty; Combination Product: VT-X7 Treatment System with Vancomycin Hydrochloride
- Control (Active Comparator): Standard of care for treatment of chronic PJI - two-stage exchange arthroplasty: surgical removal of the infected implant, aggressive debridement, and exchange arthroplasty with administration of adjuvant systemic antibiotics and temporary antibiotic-impregnated cement spacer.
  Interventions: Drug: Standard of Care; Procedure: Two-stage exchange arthroplasty

INTERVENTIONS:
Combination Product: VT-X7 Treatment System with Tobramycin Sulfate — Seven-day local antibiotic irrigation with tobramycin sulfate via the VT-X7 Knee or Hip Spacer.
  Arms: Experimental
Drug: Standard of Care — Forty-two days (minimum) systemic antibiotic administration adjuvant to two-stage exchange arthroplasty with temporary antibiotic-impregnated cement spacer per standard of care. Antibiotics will be selected by treatment provider and administered in accordance with national and local treatment guidelines.
  Arms: Control
Procedure: Two-stage exchange arthroplasty — Stage 1 consists of surgical removal of the infected prosthesis, debridement, and implantation of a temporary spacer. Stage 2 surgery consists of explantation of the temporary spacer, debridement, and implantation of a permanent prosthesis, followed by systemic administration of postoperative antibiotics for 42 days (inclusive) to 90 days (inclusive).
Combination Product: VT-X7 Treatment System with Vancomycin Hydrochloride — Seven-day local antibiotic irrigation with vancomycin hydrochloride via the VT-X7 Knee or Hip Spacer.
  Arms: Experimental

SUMMARY:
Study Type: A multi-site, parallel group, randomized trial.

Study Objectives: The objective is to evaluate safety and determine preliminary efficacy of VT-X7 (Vancomycin and Tobramycin Exchanged over 7 Days). Efficacy is evaluated as superiority of the Experimental Arm in a composite endpoint of Overall Success at 90 days, consisting of a revision prosthesis implanted at Stage 2, patient survival, absence of reoperation and absence of periprosthetic joint infection (PJI). Secondary objectives are to evaluate superiority at 365 days in a composite endpoint of Overall Success, and in separate secondary endpoints for quality of life and patient survival. The exploratory objective is to compare Experimental and Control Arms in exploratory endpoints.

Follow-up: Patients will be evaluated at 90-, 180-, and 365-day follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for two-stage exchange arthroplasty due to hip or knee PJI
* Signed informed consent
* 22 to 84 years of age (inclusive)
* Medical clearance for surgery
* Preoperative diagnosis of PJI of the hip or knee per the International Consensus Meeting of Musculoskeletal Infection 2018 definition of Periprosthetic Hip and Knee Infection

Exclusion Criteria:

* Patients with 2 or more prior one-stage or two-stage exchange arthroplasties of the infected joint;
* Patients with acute PJI, defined as total joint arthroplasty surgery within 4 weeks prior to enrollment (Stage 1) in this study;
* Patients with bacteremia or positive bacterial blood culture in the last 30 days;
* Patients with concurrent PJI of more than one joint;
* Patients with ongoing active infection of an intravenous site;
* Patients who require long-term anticoagulation or antiplatelet therapy, and for whom bridging or withholding therapy is not recommended based on the individual's clinical condition;
* Patients with advanced renal insufficiency (chronic kidney disease Stage 4 or greater or glomerular filtration rate <30 mL/min);
* Patients on chemotherapy for malignant disease;
* Patients on systemic glucocorticoid therapy (prednisone >10 mg/day or equivalent);
* Patients with immunodeficiency (e.g., splenectomy, sickle cell anemia, Stage 3 human immunodeficiency virus infection, primary immunodeficiency disease, except immunodeficiency due to immunosuppressive therapy).
* Patients who have an allergy to vancomycin hydrochloride or tobramycin sulfate (Note: prior history of red man syndrome is not considered an allergy);
* Patients who have an allergy to titanium, titanium alloys, polymethylmethacrylate or polyurethane.
* Patients who are pregnant or planning to become pregnant in the next 12 months;
* Patients in whom negative pressure wound therapy is contraindicated;
* Patients with a fungal PJI;
* Patients who have a skeletal defect greater than 150 mm in length in the tibia or femur of the infected joint;
* Patients who have a planned surgical procedure within 6 months of enrollment that can impact the conduct of the study;
* Patients who are breastfeeding at the screening visit;
* Patients who are incarcerated or are facing impending incarceration;
* Patients who have been in treatment or referred for treatment for substance abuse within the past year;
* Patients with any medical condition, including schizophrenia or another psychiatric disorder with hallucinations and/or delusions, that would interfere with the interpretation of the study results, the conduct of the study, or patient participation would not be in the best interest of the patient in the opinion of the Study Site Principal Investigator;
* Patients who will participate in another clinical study of an investigational drug or investigational device or have participated in another clinical study of an investigational drug or investigational device within the past 30 days that would interfere with the interpretation of the study results or conduct of the study;
* Patients who are judged by the Investigator to be unsuitable for the study.
* Patients receiving immunosuppressive drug therapy for bone marrow or another transplant;
* Patients currently or previously enrolled in this study;
* Patients who receive therapy including any of the following biologic agents, which will not be withheld for a period beginning at least one dosing cycle (minimum 7 days) prior to Stage 1 surgery and ending at least 14 days following Stage 2 surgery:

Adalimumab (Humira) Tocilizumab (Actemra) Etanercept (Enbrel) Anakinra (Kineret) Golimumab (Simponi) Secukinumab (Cosentyx) Infliximab (Remicade) Ustekinumab (Stelara) Abatacept (Orencia) Rituximab (Rituxan) Certolizumab (Cimzia) Tofacitinib (Xeljanz) Belimumab (Benlysta)

Ages: 22 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of Overall Success at 90 days | 90 days
  Composite endpoint of Overall Success at 90 days consisting of:
  * Stage 2 revision prosthesis implanted;
  * Absence of PJI* post-Stage 2;
  * Absence of reoperation*** of the affected joint pre- or post- Stage 2; and
  * Absence of mortality.
    * If clinical evidence of infection is present post-Stage 2 surgery, use the International Consensus Meeting on Musculoskeletal Infection 2018 guidelines for definitive PJI confirmation.
      * Reoperation includes only procedures to irrigate, debride, and remove or replace the Stage 1 spacer or any Stage 2 implant component.

SECONDARY OUTCOMES:
Composite endpoint of Overall Success at 180 days | 180 days
  Composite endpoint of Overall Success at 180 days consisting of:
  * Stage 2 revision prosthesis implanted;
  * Absence of PJI* post-Stage 2;
  * Absence of continued antibiotic therapy for treatment or prophylaxis of PJI **;
  * Absence of reoperation*** of the affected joint pre- and post-Stage 2; and
  * Absence of mortality.
    * If clinical evidence of infection is present post-Stage 2 surgery, use International Consensus Meeting on Musculoskeletal Infection 2018 guidelines for definitive PJI confirmation.
      * Continued antibiotic therapy includes antibiotic therapy at 180 days or beyond 12 weeks post-Stage 2 surgery, excluding antibiotics for documented pre-procedural prophylaxis or infection other than PJI.
        * Reoperation includes only procedures to irrigate, debride, remove or replace the Stage 1 spacer or any Stage 2 implant component.
Composite endpoint of Overall Success at 365 days consisting of: | 365 days
  Composite endpoint of Overall Success at 365 days consisting of:
  * Stage 2 revision prosthesis implanted;
  * Absence of PJI* post-Stage 2;
  * Absence of continued antibiotic therapy for treatment or prophylaxis of PJI **;
  * Absence of reoperation*** of the affected joint pre- and post-Stage 2; and
  * Absence of mortality.
    * If clinical evidence of infection is present post-Stage 2 surgery, use International Consensus Meeting on Musculoskeletal Infection 2018 guidelines for definitive PJI confirmation.
      * Continued antibiotic therapy includes antibiotic therapy at 365 days or beyond 12 weeks post-Stage 2 surgery, excluding antibiotics for documented pre-procedural prophylaxis or infection other than PJI.
        * Reoperation includes only procedures to irrigate, debride, remove or replace the Stage 1 spacer or any Stage 2 implant component.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Springer, MD, Principal Investigator — Ortho Carolina
Locations (17):
- United States (17):
  - University of Arizona, Phoenix, Phoenix, Arizona
  - Harbor-UCLA Medical Center, Torrance, California
  - VA Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Cleveland Clinic, Weston, Florida
  - University of Kentucky, Lexington, Kentucky
  - Covenant Medical Center, Saginaw, Michigan
  - New York University, New York, New York
  - Columbia, New York, New York
  - OrthoCarolina Research Institute, Inc, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Integris Southwest Medical Center, Oklahoma City, Oklahoma
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania
  - Texas Health Presbyterian, Plano, Texas
  - University of Utah, Salt Lake City, Utah
  - UVA Orthopedics Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No